CLINICAL TRIAL: NCT07214896
Title: HEALTH: Humanoid Evaluation and Learning Trial in Coalition-Aligned Healthcare Settings
Brief Title: Deployment and Evaluation of Humanoid Robotics in Coalition-Aligned Clinical Care Settings
Acronym: HEALTH
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: Truway Health, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: TRU-HUM-CLIN-2025-PRS
Record Dates: First submitted 2025-10-08; First posted 2025-10-09 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Mobility Impairment; Clinical Workflow Optimization; Sanitation Protocol Compliance; ESG-linked Healthcare Robotics Deployment
Keywords: Humanoid robotics in healthcare; Clinical deployment of humanoid robots; Biometric audit scoring; ESG compliance in clinical settings; Stem cell integration in robotics; Skin cell regeneration for humanoid units; Blockchain wage token for robotics; FX arbitrage in healthcare robotics; Coalition-aligned clinical trial; Metro-scale robotics deployment; Patient mobility assistance; Sanitation protocol automation; DAO-governed healthcare infrastructure; 1031 exchange yield farming in clinical care; Adaptive learning in humanoid systems; Public oversight of robotic healthcare trials

STUDY DESIGN:
Intervention Model Description: Humanoid robotics units are deployed across multiple metro healthcare facilities in parallel. Each facility represents a distinct intervention arm with tailored deployment protocols, biotech integration (skin/stem cell dips), and wage token logic. Outcomes are measured independently across arms using biometric audit scoring and ESG compliance metrics.
Masking Description: N/A - All stakeholders, including facility managers, auditors, and coalition observers, are aware of humanoid deployment and performance tracking.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | Unapproved Device: Yes | US Export: Yes

ARMS (4):
- New York Facility - Skin Cell Deployment (Experimental): Humanoid units deployed in patient intake and sanitation roles. Enhanced with keratinocyte-based skin cell dips to improve tactile sensitivity and surface regeneration.
  Assigned Roles: Intake assistant, sanitation technician
  Biometric Focus: Motor function, ESG compliance
  Interventions: Biological: Skin Cell Dip
- Austin Facility - Stem Cell Cognitive Enhancement (Experimental): Humanoid units deployed in mobility and R&D support roles. Enhanced with iPSC-derived stem cell dips targeting neural responsiveness and adaptive learning.
  Assigned Roles: Mobility assistant, lab technician
  Biometric Focus: Cognitive response, biotech retention
  Interventions: Biological: Stem Cell Dip
- Frankfurt Facility - ESG Optimization (Experimental): Humanoid units deployed in ESG-linked sanitation and logistics roles. Monitored for energy usage, carbon offset, and protocol adherence.
  Assigned Roles: ESG sanitation, logistics handler
  Biometric Focus: ESG compliance, human interaction
  Interventions: Behavioral: ESG Compliance Monitoring, Operational protocol
- Tokyo Facility - Wage Token Calibration (Experimental): Humanoid units deployed in public interface and intake roles. Wage tokens minted based on biometric audit scores and task completion.
  Assigned Roles: Receptionist, intake coordinator
  Biometric Focus: Wage token distribution, interaction scoring
  Interventions: Other: Wage Token Distribution

INTERVENTIONS:
Biological: Skin Cell Dip — Lab-grown keratinocyte dip applied to humanoid units to improve tactile sensitivity and surface regeneration.
  Arms: New York Facility - Skin Cell Deployment
Biological: Stem Cell Dip — iPSC-derived neuroblast dip applied to humanoid units to enhance neural responsiveness and adaptive learning.
  Arms: Austin Facility - Stem Cell Cognitive Enhancement
Other: Wage Token Distribution — HumanoidWage (HMW) tokens minted and distributed based on biometric audit scores and ESG task completion.
  Other Names: Blockchain-based compensation
  Arms: Tokyo Facility - Wage Token Calibration
Behavioral: ESG Compliance Monitoring, Operational protocol — Real-time tracking of energy usage, sanitation cycles, and carbon offset metrics via coalition dashboard.
  Arms: Frankfurt Facility - ESG Optimization

SUMMARY:
This clinical trial evaluates the deployment of humanoid robotics in coalition-aligned healthcare settings. The study measures biometric performance, ESG compliance, and operational impact across patient care, sanitation, and intake workflows. Humanoid units are enhanced via biotech integration and compensated through blockchain-based wage tokens. Outcomes will inform coalition governance, wage calibration, and metro-scale deployment strategies.

DETAILED DESCRIPTION:
The HEALTH trial (Humanoid Evaluation and Learning Trial in Healthcare) is a coalition-aligned clinical study designed to assess the deployment of humanoid robotics in real-world care environments. Conducted across metro facilities in New York, Austin, Frankfurt, and Tokyo, the trial evaluates robotic performance in patient intake, sanitation, mobility assistance, and ESG-linked operations.

Humanoid units are enhanced through biotech integration, including skin cell regeneration dips and stem cell neural augmentation. Each unit is tracked via biometric audit scoring across five dimensions: motor function, cognitive response, ESG compliance, biotech retention, and human interaction. Scores are notarized via SHA-256 and published to the coalition dashboard.

Wage tokens (HumanoidWage, HMW) are minted based on performance thresholds and distributed through smart contracts to deployed units. FX arbitrage across Tokyo and Frankfurt informs reinvestment logic and 1031 exchange-backed yield farming pools. DAO voting governs deployment, wage calibration, and protocol expansion.

This trial aims to establish scalable, transparent frameworks for humanoid integration in healthcare, anchored in coalition governance, public oversight, and metro-ready infrastructure.

ELIGIBILITY:
Inclusion Criteria:

- Age 18-75 years

Able to provide informed consent

Facility staff, clinical auditors, ESG observers, or coalition stakeholders

Willing to interact with humanoid robotics in clinical workflows

Available for biometric feedback and observational logging over 90 days

Exclusion Criteria:

- Cognitive impairment preventing informed consent

Active infectious disease requiring isolation

Prior adverse reaction to biotech-enhanced robotics

Involvement in conflicting clinical trials

Inability to comply with protocol procedures or coalition transparency requirements

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-10-06 (Actual); Primary Completion 2031-10-06 (Estimated); Study Completion 2031-10-06 (Estimated)

PRIMARY OUTCOMES:
Biometric Audit Score ≥85 Across Five Performance Dimensions | Measured at Day 30 Post-Deployment
  This outcome assesses the performance of humanoid robotics units deployed in coalition-aligned healthcare settings. Each unit is scored across five biometric dimensions: motor function, cognitive response, ESG compliance, biotech integration, and human interaction. Scores are notarized via SHA-256 and published to the coalition dashboard. Units achieving a composite score ≥85 are eligible for wage token bonuses, dip protocol expansion, and DAO-backed facility scaling.

SECONDARY OUTCOMES:
ESG Audit Compliance Score ≥90 | Humanoid units are evaluated for ESG-linked performance including energy usage, sanitation protocol adherence, and carbon offset metrics. Scores are published to the coalition dashboard and notarized via SHA-256. Units scoring ≥90 contribute to DAO-backe
  Measured at Day 60 Post-Deployment
Wage Token Distribution Volume per Unit | Continuous Monitoring Over 90 Days
  Tracks the volume of HumanoidWage (HMW) tokens minted and distributed to each humanoid unit based on biometric audit scores and task completion. Token flow is logged on-chain and used to calibrate coalition wage pools and reinvestment logic.
Clinical Workflow Efficiency Increase ≥15% | Measured at Day 90 Post-Deployment
  Assesses improvements in patient intake speed, sanitation cycle time, and mobility assistance throughput across facilities. Benchmarked against pre-deployment baselines and validated by coalition auditors.

CONTACTS AND LOCATIONS:
Overall Officials: Gavin C Solomon, President & CEO, Principal Investigator — Truway Health, Inc.
Locations (4):
- United States (2):
  - Truway Health, Inc. , View 34, 401 E 34th Street, S11P, New York, NY 10016, New York, New York
  - Coalition Retrofit Clinic - Austin, TX, Austin, Texas
- ESG Compliance Lab, Frankfurt, Germany
- Public Interface Pilot, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) collected during this trial-including biometric audit scores, ESG compliance metrics, and wage token distribution logs-will be shared with qualified researchers upon request. Data will be de-identified, SHA-256 notarized, and made available through Truway Health's coalition dashboard and secure data access portal. Access will require submission of a research proposal, DAO approval, and compliance with coalition transparency protocols.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: IPD and supporting documents will be available starting April 1, 2026, following primary study completion. Access will remain open for 5 years, until April 1, 2031, via Truway Health's secure coalition dashboard and data access portal.
Access Criteria: Qualified researchers, coalition partners, and regulatory agencies may request access to de-identified IPD, biometric scores, ESG metrics, wage token logs, and analytic code. Access requires submission of a research proposal, DAO approval, and compliance with Truway Health's transparency and data governance protocols.
URL: https://www.truwayhealth.com

REFERENCES:
- See also: health-trial — https://www.truwayhealth.com
- See also: ipd-sharing — https://www.truwayhealth.com
- See also: coalition-dashboard — https://www.truwayhealth.com
- Available data/document: Individual Participant Data Set: De-identified biometric audit — https://truwayhealth.com — truwayhealth.com
- Available data/document: Individual Participant Data Set: ESG compliance logs — https://truwayhealth.com — truwayhealth.com
- Available data/document: Individual Participant Data Set: Wage token minting and transfe — https://truwayhealth.com — truwayhealth.com
- Available data/document: Individual Participant Data Set: SHA-256 notarized study protoc — https://www.truwayhealth.com — truwayhealth.com
- Available data/document: Individual Participant Data Set: Statistical analysis plan (SAP — https://www.truwayhealth.com — truwayhealth.com
- Available data/document: Individual Participant Data Set: Informed consent form (ICF) — https://www.truwayhealth.com — truwayhealth.com
- Available data/document: Individual Participant Data Set: Clinical study report (CSR) — https://www.truwayhealth.com — truwayhealth.com
- Available data/document: Individual Participant Data Set: Analytic code for biometric sc — https://www.truwayhealth.com — truwayhealth.com